CLINICAL TRIAL: NCT03000452
Title: MEDI4736-MM-005 (FUSION MM-005): A Phase 2, Multicenter, Single-Arm, Study to Determine the Efficacy for the Combination of Durvalumab (DURVA) Plus Daratumumab (DARA) (D2) in Subjects With Relapsed and Refractory Multiple Myeloma (RRMM) That Have Progressed While on Current Treatment Regimen Containing Daratumumab.
Brief Title: A Study to Determine the Efficacy of the Combination of Daratumumab (DARA) Plus Durvalumab (DURVA) (D2) in Subjects With Relapsed and Refractory Multiple Myeloma (RRMM)
Acronym: FUSION-MM-005
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MEDI4736-MM-005
Record Dates: First submitted 2016-12-19; First posted 2016-12-22 (Estimated); Results first posted 2018-10-16 (Actual); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; Daratumumab; Durvalumab; Relapsed and Refractory Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — daratumumab; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Administration of Daratumumab (DARA) plus Durvalumab (DURVA) (Experimental): Subjects will also receive IV DURVA at 1500 mg on Day 2 (Cycle 1) and on Day 1 (Cycles ≥ 2) of each 28-day treatment cycle.
  Subjects will receive intravenous (IV) DARA at 16 mg/kg on the same dosing schedule (weekly [QW], every 2 weeks [Q2W], or every 4 weeks [Q4W] of each 28-day treatment cycle) received during their last prior therapy containing DARA at the time of DARA progression
  Interventions: Drug: DARATUMUMAB; Drug: DURVALUMAB

INTERVENTIONS:
Drug: DARATUMUMAB — DARATUMUMAB
  Other Names: DARA
Drug: DURVALUMAB — DURVALUMAB
  Other Names: MEDI4736; DURVA

SUMMARY:
This is a single-arm, multicenter, Phase 2 study to evaluate the efficacy and safety of the combination regimen of daratumumab plus durvalumab (D2). The study will consist of 2 parts; Part 1 has a 2-stage design while Part 2 consists of an expansion phase. Subjects will receive intravenous (IV) DARA at 16 mg/kg on the same dosing schedule (weekly [QW], every 2 weeks [Q2W] or every 4 weeks [Q4W] of each 28-day cycle) received on their last prior therapy containing DARA. The dosing schedule for DARA may be adjusted during the course of the study as outlined in the protocol. Subjects will also receive IV DURVA at 1500 mg on Day 2 (Cycle 1) and on Day 1 (Cycles ≥ 2) of each 28-day treatment cycle.

DETAILED DESCRIPTION:
Indication:

This study will include subjects that have relapsed and refractory multiple myeloma (RRMM) after treatment with at least 3 prior antimyeloma therapies, including a proteasome inhibitor (PI) and an immunomodulatory drug (IMiD®) or after development of double-refractoriness to a both a PI and an IMiD.

The most recent multiple myeloma (MM) treatment regimen should contain daratumumab (DARA) and subjects must have progressed on DARA while on this regimen. Stage 1 A cohort of 18 subjects will be enrolled to determine the preliminary efficacy of DARA plus DURVA. Once the 18 subjects have been enrolled, an interim analysis for futility purpose will be conducted to determine if the study can proceed to Stage 2.

Early Safety Monitoring Once 6 subjects have been enrolled and completed the first treatment cycle in Stage 1 of this study, the enrollment continuity would depend on the availability of safety data from the on-going Phase 2 study (MEDI4736-MM-003) of DARA and DURVA in previously DARA-naïve patients.

* If MEDI4736-MM-003 safety data are available and the tolerability profile of DARA plus DURVA has been determined to be adequate, then enrollment will continue as planned in Stage 1 without an early safety monitoring review of the data.
* If safety data are not available enrollment in this study will be paused for a review of the safety profile of DARA plus DURVA by a Dose Review Team (DRT), using the data from the first 6 patients.
* If ≥ 1 of the first 6 patients experiences a dose-limiting toxicity (DLT), the study will be halted for review and a change in the dosing regimen may be implemented.
* The DRT will consist of the Celgene Medical Monitor, Celgene lead Safety Physician, Celgene biostatistician, other Celgene functional area representatives, as appropriate, study specific consultants (MD/PhD), and site investigator and/or designees who have enrolled subjects to the study.
* All available safety and, if applicable, PK/(pharmacodynamic) Pd, biomarker, and preliminary efficacy data will be reviewed and can be considered in the DRT's decisions.
* A DRT meeting will be held to review all data and make decisions regarding continuity of the study.

Dose-limiting Toxicity

Dose-limiting toxicities (DLTs) may be evaluated during the DLT evaluation period for the initial 6 patients in Part 1 of the study. The DLT evaluation period will be defined as the first treatment cycle. Subjects are considered evaluable for assessment of DLT if they:

* Receive at least 1 dose of study treatments and experience a DLT OR
* Receive 1 dose of DURVA, 4 doses of DARA and complete the safety follow-up through the end of the DLT evaluation period.

Grading of DLTs will be according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 4.03.

A DLT will be defined as below:

Hematologic DLT

1. Grade 4 neutropenia observed for greater than 5 days duration
2. Grade 3 neutropenia associated with fever (≥ 38.5 °C) of any duration.
3. Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding, or any requirement for platelets transfusion.
4. Any other Grade 4 hematologic toxicity that does not resolve to subject's pretreatment baseline level within 72 hours
5. Grade 4 anemia, unexplained by underlying disease. Non-hematologic DLT

a. Any nonhematological toxicity ≥ Grade 3 except for alopecia and nausea controlled by medical management b. Any treatment interruption greater than 2 weeks due to an AE. While the rules for adjudicating DLTs in the context of dose escalation are specified above, an AE not listed above may be defined as a DLT after consultation with the Sponsor and investigators, based on the emerging safety profile.

Stage 2 If 3 or more subjects achieved a response (PR or better) out of the 18 subjects at the end of Stage 1, an additional 32 subjects will be enrolled to evaluate the safety and efficacy of DARA plus DURVA.

Part 2: Expansion Upon completion of Part 1, if at least 9 subjects achieve a response (PR or better) out of a total of 50 subjects and it is determined to further confirm the efficacy and safety of DARA plus DURVA, an additional 70 subjects may be enrolled.

An Independent Response Adjudication Committee (IRAC) will be set up for this trial to review study data. The IRAC will determine tumor response to therapy and to confirm the time of disease progression (PD) (if disease progressed) at scheduled or unscheduled visits for each subject.

The safety and efficacy of the study will be monitored by an independent Data Monitoring Committee (DMC) who are not involved in the trial conduct. The DMC will meet up and review study data at pre specified intervals throughout the trial.

In the event that the trial is halted for early safety monitoring, evaluation of the emerging safety data from the initial 6 patients enrolled in Part 1 will be performed by the Dose Review Team (DRT).

Safety data will be monitored by the Celgene Medical Monitor and Safety Physician on an ongoing basis throughout the study. Should a significant safety issue be identified, the DMC will be convened to make a recommendation as to the future conduct of the study.

The decision to discontinue a subject, which will not be delayed or refused by the Sponsor, remains the responsibility of the treating physician. However, prior to discontinuing a subject, the Investigator may contact the Medical Monitor and forward appropriate supporting documents for review and discussion.

The study will be conducted in compliance with the International Council on Harmonisation (ICH) of Technical Requirements for Registration of Pharmaceuticals for Human Use/Good Clinical Practice (GCP) and applicable regulatory requirements.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject received at least 3 prior anti-myeloma regimens including a proteasome inhibitor (PI) and an immunomodulatory agent or is double-refractory to a PI and an immunomodulatory agent.

   * Induction, bone marrow transplant with or without maintenance therapy is considered one regimen.
   * Refractory is defined as disease that is nonresponsive on therapy, or progresses within 60 days of last therapy. Nonresponsive disease is defined as either failure to achieve minimal response or development of progressive disease while on therapy.
   * For subjects who received more than 1 regimen containing a PI their disease must be refractory to the most recent PI containing regimen.
   * For subjects who received more than 1 regimen containing a immunomodulatory agent their disease must be refractory to the most recent immunomodulatory agent containing regimen.
2. All subjects must have failed Daratumumab (DARA) either as a single agent or in combination on last Multiple myeloma (MM) therapy. Failure is defined as disease progression(PD) on DARA either as a single agent or in combination.
3. Subject has measurable disease defined as:

   1. M-protein (serum protein electrophoresis (sPEP) or urine protein electrophoresis (uPEP): sPEP ≥ 0.5 g/dL or uPEP ≥ 200 mg/24 hours) and/or
   2. Light chain MM without measurable disease in the serum or the urine: serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa lambda free light chain ratio
4. Subject achieved a response (minimal response [MR] or better) to at least 1 prior treatment regimen.
5. Subject has an Eastern Cooperative Oncology Group (ECOG) Performance Status score of 2 or less.
6. Subject's toxicities resulting from previous therapy (including peripheral neuropathy) have resolved or stabilized to ≤ Grade 1.
7. Subject is at least 18 years of age the time of signing the informed consent form (ICF).
8. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
9. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
10. Females of childbearing potential (FCBP) must:

    a. Have 2 negative pregnancy tests as verified by the investigator prior to starting study treatment. This applies even if the subject practices true abstinence from heterosexual contact.

    i. Negative serum pregnancy test at screening ii. Negative serum or urine pregnancy test (investigator's discretion) within 72 hours prior to starting study treatment (Cycle 1, Day 1), and before beginning each subsequent cycle of treatment, and after end of study treatment.

    b. Either practice true abstinence from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, effective contraception without interruption (eg, oral, inject able, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; true abstinence; or vasectomized partner), 28 days prior to starting study treatment, during the study therapy (including dose interruptions), and for at least 90 days after discontinuation of study treatment.

    c. Agree to abstain from breastfeeding during study participation and for at least 90 days after the last dose of Daratumumab (DARA) or Durvalumab (DURVA), whichever is later.

    d. Refrain from egg cell donation for at least 90 days after the final dose of DURVA or DARA, whichever is later.
11. Male subjects must:

    1. Either practice true abstinence (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 90 days following study treatment discontinuation, even if he has undergone a successful vasectomy.
    2. Refrain from sperm donation for at least 90 days after the final dose of DURVA or DARA, whichever is later.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has had prior exposure to anti-CTLA-4, anti-PD-1 (Programmed cell death-1), anti-PD-L1 (Programmed death-ligand 1) Monoclonal antibody (mAbs), or cancer vaccines
2. Subject has received autologous stem cell transplantation (ASCT) within 12 weeks before the date of randomization.
3. History of organ or allogeneic stem cell transplantation
4. Subject received any of the following within the last 14 days of initiating study treatment:

   1. Plasmapheresis
   2. Major surgery (as defined by the investigator)
   3. Radiation therapy other than local therapy for myeloma associated bone lesions
   4. Use of any systemic anti-myeloma drug therapy (except for DARA either alone or in combination with other agents given with it)
5. Subject received prior treatment with a monoclonal antibody within 5 half-lives of initiating study treatment, other than DARA.
6. Subject is receiving concurrent chemotherapy or biologic or hormonal therapy for cancer treatment. Note: Concurrent use of hormones for noncancer-related conditions (eg, insulin for diabetes and hormone replacement therapy) is acceptable.
7. Subject has any of the following laboratory abnormalities:

   1. Absolute neutrophil count (ANC) < 1,000/µL
   2. Platelet count: < 75,000/µL (it is not permissible to transfuse a subject to reach this level)
   3. Hemoglobin < 8 g/dL (< 4.9 mmol/L) (it is not permissible to transfuse a subject to reach this level)
   4. Creatinine clearance (CrCl) < 45 mL/min (calculated using the Cockcroft-Gault formula or directly calculated from the 24-hour urine collection method)
   5. Corrected serum calcium > 13.5 mg/dL (> 3.4 mmol/L)
   6. Serum aspartate aminotransferase (AST) or alanine aminotransferase (ALT) > 2.5 × upper limit of normal (ULN)
   7. Serum total bilirubin > 1.5 × upper limit of normal (ULN) or > 3.0 mg/dL for subjects with documented Gilbert's syndrome
8. Subject has clinical evidence of central nervous system (CNS) or pulmonary leukostasis, disseminated intravascular coagulation, or CNS MM
9. Subject has known chronic obstructive pulmonary disease (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Note that forced expiratory testing (FEV1) is required for subjects suspected of having COPD and subjects must be excluded if FEV1 is < 50% of predicted normal.
10. Subject has known moderate or severe persistent asthma within the past 2 years or uncontrolled asthma of any classification. Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.
11. Subject has plasma cell leukemia, Waldenstrom's macroglobulinemia, POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes), or amyloidosis
12. Subject has nonsecretory MM
13. Subject has known allergy or hypersensitivity to study drug formulations
14. Subject has active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [eg, colitis, Crohn's disease], diverticulitis, celiac disease, irritable bowel disease, or other serious gastrointestinal chronic conditions associated with diarrhea; systemic lupus erythematosus; Wegener syndrome; myasthenia gravis; Graves' disease; rheumatoid arthritis, hypophysitis, uveitis, etc) within the past 3 years prior to the start of treatment. The following are exceptions to this criterion:

    1. Subjects with vitiligo or alopecia.
    2. Subjects with hypothyroidism (eg, following Hashimoto's disease) stable on hormone replacement.
    3. Psoriasis not requiring systemic treatment.
15. Subject has history of primary immunodeficiency
16. Subject is positive for human immunodeficiency virus (HIV-1), chronic or active hepatitis B or active hepatitis A or C.
17. Subject has received live, attenuated vaccine within 30 days prior to the first dose of DURVA (NOTE: Subjects, if enrolled, should not receive live vaccine during the study and through 30 days after the last dose of DURVA)
18. Subject is currently using or has used immunosuppressive medication within 14 days prior to the first study dose of study treatment. The following are exceptions to this criterion:

    1. Intranasal, topical, inhaled, or local steroid injections (eg, intra-articular injection).
    2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent.
    3. Steroids as premedication for hypersensitivity reactions (eg, infusion-related reactions, computed tomography [CT] scan premedication).
19. Subject has any one of the following:

    1. Clinically significant abnormal Electrocardiogram (ECG) finding at screening
    2. Congestive heart failure (New York Heart Association Class III or IV)
    3. Myocardial infarction within 12 months prior to starting study treatment
    4. Unstable or poorly controlled angina pectoris, including Prinzmetal variant angina pectoris
20. Subject has prior history of malignancies, other than MM, unless the subject has been free of the disease for ≥ 5 years with the exception of the following noninvasive malignancies:

    1. Basal cell carcinoma of the skin
    2. Squamous cell carcinoma of the skin
    3. Carcinoma in situ of the cervix
    4. Carcinoma in situ of the breast
    5. Incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is curative
21. Subject is a female who is pregnant, nursing, or breastfeeding, or who intends to become pregnant during the participation in the study.
22. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
23. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
24. Subject has any condition that confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-03-14 (Actual); Primary Completion 2017-09-18 (Actual); Study Completion 2017-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Novick, MD, PhD, Study Director — Celgene Corporation
Locations (25):
- United States (12):
  - City of Hope Cancer Center, Duarte, California
  - Cancer Center of Central Connecticut, Southington, Connecticut
  - Parkview Research Center, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - University of Kansas Hospital, Westwood, Kansas
  - University of Maryland School of Med, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - John Theurer Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - Morristown Memorial Hosp, Morristown, New Jersey
  - OHSU, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
- Austria (3):
  - Universitaetsklinik Innsbruck, Innsbruck
  - Salzburger Landkliniken St. Johanns-Spital, Salzburg
  - Medizinische Universitat Wien, Vienna
- Alexandra General Hospital of Athens, Athens, Greece
- UMCU Utrecht, Utrecht, Netherlands
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol Can Ruti, Badalona (Barcelona)
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Universitario Dr. Pesset, Valencia
- Sweden (4):
  - Falu lasarett, Falun SE
  - Helsingborg hospital, Helsingborg
  - Lund University Hosptial, Lund
  - Karolinska University Hospital Huddinge, Stockholm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 8 sites in 4 countries including Greece, Spain, Sweden and the United States, from 14 March 2017 to 04 December 2017
Pre-assignment Details: Eligible participants included those with relapsed and refractory multiple myeloma (RRMM) who progressed on daratumumab (DARA) while on a DARA-containing regimen as the most recent multiple myeloma (MM) therapy. Participants had to have received at least 3 prior anti-myeloma therapies.
Groups:
- Daratumumab and Durvalumab: Participants received intravenous daratumumab at 16 mg/kg on the same dosing schedule (weekly, every 2 weeks, or every 4 weeks of each 28-day treatment cycle) on their last prior therapy containing daratumumab regimen. The dosing schedule for daratumumab could be adjusted during the course of the study, provided the participant had a response of stable disease or better. Participants also received IV durvalumab at 1500 mg on Day 2 of Cycle 1 and then on Day 1 of Cycles ≥ 2 of each 28-day treatment cycle. Participants could continue on study treatment until progressive disease or unacceptable toxicity.
Period: Treatment Period
Arm/Group | Daratumumab and Durvalumab
Started | 18
Completed | 0
Not Completed | 18
Not completed — Death | 1
Not completed — Progressive Disease (PD) | 14
Not completed — Physician Decision | 1
Not completed — Miscellaneous | 2
Period: Follow-Up Period
Arm/Group | Daratumumab and Durvalumab
Started | 17 (1 participant died in Cycle 1 due to PD prior to evaluation.)
Completed | 10
Not Completed | 7
Not completed — Study Terminated by Sponsor | 1
Not completed — Death | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Population = all participants who enrolled in the study.
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.8 (11.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 7
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Black or African American | 1
  White | 15
  Not Collected or Reported | 2
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — ECOG PS is used by physicians and researchers to assess how a subject's disease is progressing, and how the disease affects the daily living activities and determine appropriate treatment and prognosis. 0 = Fully Active, able to carry on all pre-disease performance without restriction; 1 = Restricted, in physically strenuous activity but ambulatory; 2 = Ambulatory and capable of all self-care; unable to carry out work activities. 3 = Capable of only limited self-care, confined to bed or chair >50% of waking hours 4 = Completely Disabled, cannot carry on any self-care 5 = Dead
  Participants
    0 = Fully Active | 12
    1 = Restrictive but ambulatory | 5
    2 = Ambulatory but unable to work | 1
    3 = Limited Self-Care | 0
International Staging System Multiple Myeloma Stage at Entry [Count of Participants; unit: Participants] — The International Staging System divides myeloma into 3 stages based only on the serum beta-2 microglobulin and serum albumin levels. Stage I: Serum beta-2 microglobulin is less than 3.5 (mg/L) and the albumin level is above 3.5 (g/L); Stage II: Neither stage I or III, meaning that either: # The beta-2 microglobulin level is between 3.5 and 5.5 (with any albumin level), OR # The albumin is below 3.5 while the beta-2 microglobulin is less than 3.5 Stage III: Serum beta-2 microglobulin is greater than 5.5.
  Participants
    Stage I | 5
    Stage II | 4
    Stage III | 9
    Missing | 0
Number of Prior Regimens [Median (Full Range); unit: Regimens] | 4.5 [3 to 16]

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Objective Response According to International Myeloma Working Group (IMWG) Uniform Response Criteria
Description: Objective response is defined as a best overall response of stringent complete response (sCR), complete response (CR), very good partial response (VGPR) or partial response (PR) based on the investigator assessment: sCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤ 5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥ 90% reduction in serum M-protein and urine M-protein level < 100 mg/24 hours; PR: ≥ 50% reduction of serum M-Protein and reduction in urinary M-protein by ≥ 90% or to < 200 mg/24 hours. In addition to the above, if present at baseline a ≥ 50% reduction in the size of soft tissue plasmacytomas is also required.
Time Frame: From randomization until the data cut-off date of 17 April 2018. The median duration of treatment for durvalumab and daratumumab was 7.9 weeks and 8.0 weeks respectively.
Population: Full Analysis Set = all participants who enrolled in the study.
Measure: Number; unit: percentage of participants
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 18
percentage of participants | 0.0

2. Secondary Outcome: Time-to-Response (TTR)
Description: Time-to-response was defined as the time from treatment initiation to the first documentation of response (PR or greater) based on IMWG criteria. sCR: CR and normal free light chain (FLC) ratio and no clonal cells in bone marrow; CR: Negative serum and urine on immunofixation, disappearance of any soft tissue plasmacytomas and ≤5% plasma cells in bone marrow; VGPR: Serum and urine M-protein detectable by immunofixation but not on electrophoresis or ≥90% reduction in serum M-protein and urine M-protein level <100 mg/24 hours; PR: ≥50% reduction of serum M-Protein and reduction in urinary M-protein by ≥90% or to <200 mg/24 hours. A ≥50% decrease in the difference between involved and uninvolved FLC levels in place of the M-protein criteria or a ≥50% reduction in plasma cells in place of M-protein if baseline was ≥30%. If present at baseline a ≥50% reduction in size of soft tissue plasmacytomas.
Time Frame: as for outcome 1
Population: Analyses was not conducted for TTR due to no participant achieving a best response better than stable disease in Stage 1 of the study. Following the review of the data by the data monitoring committee (DMC) the sponsor decided to close the study as the number of responses was not reached.
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of Response (DOR)
Description: Duration of response was defined as time from the first documentation of response (PR or greater) to the first documentation of PD or death, whichever is earlier, based on the investigator assessments according to the IMWG Uniform Response Criteria.
Time Frame: as for outcome 1
Population: Analyses was not conducted for duration of response because no participant achieved a best response better than stable disease in Stage 1 of the study. Following the review of the data by the data monitoring committee the sponsor decided to close the study as the number of responses was not reached.
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival was defined as the time from treatment initiation to the first documentation of PD or death from any cause during study, whichever occurred earlier. Time to event analysis for PFS and was not analyzed due to insufficient follow up time because of early termination of the trial.
Time Frame: as for outcome 1
Population: Analyses was not conducted for PFS because no participant achieved a best response better than stable disease in Stage 1 of the study. Following the review of the data by the data monitoring committee the sponsor decided to close the study as the number of responses were not reached.
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Overall Survival was defined as the time from treatment initiation to death due to any cause. Time to event analysis for overall survival was not analyzed due to insufficient follow up time because of early termination of the trial.
Time Frame: as for outcome 1
Population: Analyses was not conducted for overall survival because no participant achieved a best response better than stable disease in Stage 1 of the study. Following the review of the data by the data monitoring committee the sponsor decided to close the study as the number of responses was not reached.
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 0

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration Of Durvalumab
Description: Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration, calculated by linear trapezoidal method when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.
Time Frame: Pharmacokinetic samples were drawn on Cycle 1 on Day 2 (C1D2) pre-dose, at the end of the infusion, on Day 8 at 144 hour post dose, on Day 15 at 312 hours post dose and on Day 22 at 480 hours post C1D2 infusion.
Population: The pharmacokinetic population included participants who received at least 1 dose of study medication and had evaluable plasma PK durvalumab profiles.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/L
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 14
day*μg/L | 3145469.40 (43.3)

7. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to Extrapolated to Infinity (AUC-inf) of Durvalumab
Description: Area under the plasma concentration-time curve from time 0 extrapolated to infinity, calculated as [AUCt + Ct/ λz]. Ct is the last quantifiable concentration. No AUC extrapolation was performed with unreliable λz. If AUC %Extrap was ≥25%, AUC inf was not reported.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/L
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 10
day*μg/L | 5634957.81 (86.8)

8. Secondary Outcome: Maximum Observed Concentration (Cmax) Of Durvalumab
Description: Maximum observed plasma concentration, obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/L
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 14
μg/L | 349391.46 (32.2)

9. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Durvalumab
Description: Time to Cmax, obtained directly from the observed concentration versus time data.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 14
days | 0.0476 [0.003 to 0.058]

10. Secondary Outcome: Terminal Half-Life (T1/2) of of Durvalumab
Description: Terminal phase half-life in plasma, calculated as [(ln 2)/λz]. t1/2 was only calculated when a reliable estimate for λz could be obtained.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: days
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 10
days | 15.71 (75.4)

11. Secondary Outcome: Apparent Total Clearance (CL/F) of of Durvalumab
Description: Apparent total clearance, calculated as [Dose/AUCinf].
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 10
L/day | 0.27 (86.8)

12. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Durvalumab
Description: Apparent volume of distribution, calculated as [(CL/F)/λz].
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 10
Liters | 5.48 (25.1)

13. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: TEAEs include AEs between the earliest of the first dose date of either study drug and 90 days after the last dose of either study drug. In addition, an AE that occurred beyond the timeframe and was assessed by the doctor as possibly related to IP was considered to be treatment-emergent. Severity was assessed using National Cancer Institute Common Toxicity Terminology Criteria for AEs (NCI CTCAE) version 4.03, where 1= Mild; 2= Moderate; 3= Severe; 4= Life-threatening; 5= Death related to AE. Serious AEs resulted in death, were life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, congenital anomaly, or resulted in a medical event that may have jeopardized the patient or required medical or surgical intervention to prevent one of the outcomes above.
Time Frame: From the date of the first dose of study drug until 90 days after the last dose of durvalumab or daratumumab , whichever is later. Maximum overall time on treatment was 16 weeks for daratumumab and durvalumab
Population: The safety population consisted of all participants who received at least one dose of Durvalumab (Durva) or Daratumumab (Dara).
Measure: Count of Participants; unit: Participants
Arm/Group | Daratumumab and Durvalumab
Number analyzed (Participants) | 18
Participants
  TEAE | 18
  TEAE Related to Durva | 1
  TEAE Related to Dara | 4
  TEAE Related to Durva or Dara | 4
  TEAE with CTCAE Grade (Gr) 3-4 | 11
  TEAE with CTCAE Grade 3-4 Related to Durva | 1
  TEAE with CTCAE Grade 3-4 Related to Dara | 2
  TEAE with CTCAE Gr 3-4 Related to Durva or Dara | 2
  TEAE with CTCAE Grade 5 | 4
  TEAE with CTCAE Grade 5 Related to Durva | 0
  TEAE with CTCAE Grade 5 Related to Dara | 0
  TEAE with CTCAE Gr 5 Related to Durva or Dara | 0
  Serious AE | 7
  Serious AE Related to Durva | 0
  Serious AE Related to Dara | 0
  Serious AE Related to Durva or Dara | 0
  TEAE leading to Interruption of Durva | 1
  TEAE leading to Interruption of Dara | 1
  TEAE leading to Interruption of Durva or Dara | 1
  TEAE interruption of Durva-without infusion delay | 1
  TEAE interruption of Dara-without infusion delay | 1

ADVERSE EVENTS:
Time Frame: From first dose of study drug to 90 days after the last dose of daratumumab and durvalumab, whichever was later, as well as SAEs made known to the investigator at any time thereafter that are suspected of being related to daratumumab or durvalumab. Maximum overall time on treatment was 16 weeks for daratumumab and durvalumab
Arm/Group | Daratumumab and Durvalumab
All-Cause Mortality (participants affected / at risk) | 4/18
Serious Adverse Events (participants affected / at risk) | 7/18
Other Adverse Events (participants affected / at risk) | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab and Durvalumab (N=18)
Cardiac failure (Cardiac disorders) | 1
General physical health deterioration (General disorders) | 4
Pyrexia (General disorders) | 1
Pneumonia (Infections and infestations) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Daratumumab and Durvalumab (N=18)
Anaemia (Blood and lymphatic system disorders) | 12
Lymphopenia (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 7
Tachycardia (Cardiac disorders) | 1
Cataract (Eye disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Chest discomfort (General disorders) | 1
Fatigue (General disorders) | 9
General physical health deterioration (General disorders) | 2
Localised oedema (General disorders) | 1
Oedema peripheral (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Herpes zoster (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Viral upper respiratory tract infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 1
Amylase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 6
Blood fibrinogen decreased (Investigations) | 1
Lipase increased (Investigations) | 1
Weight decreased (Investigations) | 3
Decreased appetite (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 3
Hyponatraemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Neuralgia (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Disorientation (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Catarrh (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Hypertension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
An independent DMC reviewed data from Part 1 Stage 1 of the study on 26 Oct 2017; based on their recommendations, Celgene decided to close the study due to unfavorable efficacy results (number of responses to move to Stage 2 was not reached).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Results from a center cannot be submitted for publication before results of multicenter study are published unless it is > 1 year since study completion. Then, Investigator can publish if manuscript is submitted to Celgene 60 days prior to submission. If Celgene decides publication would hinder drug development, Investigator must delay submission for up to 90 additional days. Investigator must delete confidential information before submission and defer publication to permit patent applications.

DOCUMENTS (2):
  • Study Protocol (2016-10-03): https://cdn.clinicaltrials.gov/large-docs/52/NCT03000452/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-09): https://cdn.clinicaltrials.gov/large-docs/52/NCT03000452/SAP_001.pdf